CLINICAL TRIAL: NCT01922310
Title: Communication With Families Regarding Organ and Tissue Donation After Death in Intensive Care Study
Brief Title: Communication Regarding Organ and Tissue Donation in Intensive Care
Acronym: COMFORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NSW Organ and Tissue Donation Service (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Health Services Research
Other Study IDs: DR-01-2012; ACTRN12613000815763 (Registry Identifier: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2013-08-10; First posted 2013-08-14 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Tissue and Organ Procurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Communication intervention (Other): This study uses a single arm design with current 'controls' to explore an intervention, the procedure for providing information and requesting consent for donation, that uses new agreed best practice procedures led by specially trained intensive care health professionals. The study intervention is a staff education and training module intended to provide a framework and preparation for select critical care staff to conduct organ donation discussions in line with best practice.
  Interventions: Behavioral: Communication intervention

INTERVENTIONS:
Behavioral: Communication intervention — The intervention is a modification of current standard practice procedures for requesting consent for donation.
  The intervention period commences when the possibility of organ donation is first raised with the family, and includes the time for families to make a decision. This time may last up to 72 hours.

SUMMARY:
The overarching aim of this study is to examine the process of organ donation decision-making and to determine whether changes in requesting practices change rates of consent for donation, and other family-based outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Donation events identified by a patient who is a potential organ and tissue donor in a participating ICU or under the care of ICU health professionals.
* For the primary endpoint only, patients must not have registered their donation wishes.

Exclusion Criteria:

* A patient who is not medically suitable for organ or tissue donation.
* A patient who does not have next of kin available to participate in donation conversations.
* A patient in the ICU who is able to provide first person consent for deceased donation, for example a patient with spinal injuries.
* A patient who is suitable to donate only tissue after death.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-07-08 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Proportion of families providing consent for deceased organ donation. | Up to 72 hours subsequent to raising deceased donation with next of kin.
  Final decision of either written or verbal consent or decline to deceased organ donation provided at the hospital.

SECONDARY OUTCOMES:
Proportion of senior next of kin who report they regretted their final decision either to consent or to decline donation. | 90 days post enrollment.
  This outcome will be assesed using a telephone follow-up call.

OTHER OUTCOMES:
Health professionals' adherence rates to core elements of the intervention. | Up to 72 hours subsequent to next of kin making their final donation decision.
  This will be measured by observation and self-report at the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Herkes, Principal Investigator — NSW Organ and Tissue Donation Service
Locations (10):
- Australia (10):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - NSW Organ and Tissue Donation Service, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales

REFERENCES:
- [Derived] Potter JE, Perry L, Elliott RM, Aneman A, Brieva JL, Cavazzoni E, Cheng AT, O'Leary MJ, Seppelt IM, Herkes RG; COMFORT study investigators. Communication with Families Regarding Organ and Tissue Donation after Death in Intensive Care (COMFORT): a multicentre before-and-after study. Crit Care Resusc. 2018 Dec;20(4):268-276. PMID 30482134
- [Derived] Potter JE, Herkes RG, Perry L, Elliott RM, Aneman A, Brieva JL, Cavazzoni E, Cheng AT, O'Leary MJ, Seppelt IM, Gebski V; COMFORT study investigators. COMmunication with Families regarding ORgan and Tissue donation after death in intensive care (COMFORT): protocol for an intervention study. BMC Health Serv Res. 2017 Jan 17;17(1):42. doi: 10.1186/s12913-016-1964-7. PMID 28095838